CLINICAL TRIAL: NCT02434068
Title: Assessment of Flexible Ureteroscopy Residual Fragments
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: 11851
Record Dates: First submitted 2015-02-19; First posted 2015-05-05 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Calculi
Keywords: kidney calculi; followup studies
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stone residuals: all patients are going to be submitted to the same intervention: CT, US, KUB
  Interventions: Other: CT

INTERVENTIONS:
Other: CT — followup
  Other Names: US; KUB

SUMMARY:
Residual fragments of urinary calculi after flexible ureteroscopy (URF) can cause symptoms and additional surgeries. The assessment of residual fragments by imaging is not standardized. Computed tomography (CT) is the best way for evaluation of urinary stones, however, ionizing radiation from CT is deleterious. The aim of this study is to define which patients may avoid CT for evaluation of residual fragments after URF. 115 patients with > 18 years old undergoing URF for kidney stone < 20 mm or < 15 mm in the lower calyx diagnosed by CT will be studied. The clinical evaluation of patients will be held by the same urologist in pre-operative consultation, 7 days after the procedure, 30 days after the procedure and 100 days after the procedure. The assessment of residual fragments will be made through TC, ultrasound and Kidney-bladder-ureter KUB 90 days after the procedure. The image methods for residual fragments assessment will be compared by Cochran Test and prediction of parameters to avoid CT will be made by multiple logistic regression, using IPSS 16.0, with significant level of 5%.

DETAILED DESCRIPTION:
Flexible ureteroscopy (URF) is being widely used for the treatment of kidney stones up to 20 mm. The assessment of residual fragments must be done because they could cause pain and additional surgical interventions. However, nor the timing or modality of image study for this assessment is standardized yet.

Computed Tomography (CT) has become the standard for diagnosing urinary stones. Stone-former patients are submitted to many CT studies during life due to stone-related events. However, the cumulative exposure to the ionizing radiation of CT may induce tumors. Therefore, efforts to reduce radiation exposure are recommended such as better selection of the timing to submit the patient to CT, low radiation dose protocols and restriction of body region to be examined.

Up to 38% of the patients have residual fragments more than 2 mm assessed by CT after URF. The investigators goal is to predict witch patients should be submitted to CT for the assessment of residual fragments after URF and to evaluate the clinical significance of residual fragments and URF complications.

Method

115 consecutive symptomatic adult (>18 years-old) patients diagnosed by CT with kidney stone more than 5 mm and less than 20 mm or less than 15 mm in inferior calyx are going to be submitted to URF. Residual fragments are going to be assessed by CT, ultrasound and plain radiography during post-operative period. The study protocol is approved by our hospital's ethics committee, and written informed consent is going to be obtained from all patients according to the Declaration of Helsinki Ethical Principles for Medical Research Involving Human Subjects.

Sample size

Sample size was calculated based on the percentage of patients with residual fragments more than 2 mm by CT of 38% and by plain radiography of 17%. Therefore, sample size for a bicaudal test with significance level of 5% and test power of 95% is 115 subjects.

Exclusion factors

Patients with kidney malformations, ureteral stenosis, previous ipsilateral kidney surgery, hydronephrosis, indwelling double J stent and contraindications for URF are going to be excluded.

Flexible ureteroscopy

The procedure is going to be performed in a radiation proof operating room under general anesthesia.

A pyelography is obtained and a Nitinol 0.035" guidewire and a PTFE 0.035" guidewire are inserted up to the renal pelvis under radioscopy guidance.

Semi-rigid ureteroscopy is performed for active dilation of the ureter. Ureteral sheath 10/12F x 35 cm is than placed up to the upper ureter and the flexible ureteroscope is inserted through the ureteral sheath for direct identification of all renal calices and kidney stones before lithotripsy.

Laser lithotripsy will be performed with a 200-270 micron Holmium laser fiber until complete stone dusting or basketing of stone fragments > 2 mm with < 1.9 F tipless basket. Stone fragments < 2 mm are acceptable. Pyelography through ureteral sheath will be done to search for perforation of the urinary tract and to help proper positioning of 6 F double J stent in the renal pelvis. The ureteral sheath is going to be removed under direct ureteroscopic vision to care for ureteral lesions and ureteral stone fragments.

Follow-up

The clinical evaluation will be held by the same urologist in pre-operative consultation, 7 days after the procedure, 30 days after the procedure and 100 days after the procedure. The assessment of residual fragments will bem ade through CT, urinary tract Ultrasound (US) and X-Ray of the abdomen (Rx) in 90 days postoperatively in all patients. After the procedure, patients receive guidelines and prescribing for household use standardized pain control.

Evaluated parameters

The parameters evaluated in each patient will be: demographic data like gender, age, race, body mass index, waist circumference, kidney stone size with 3 measures diameters for calculation of maximum diameter, area and volume, measured in Hounsfield units of kidney stone, number of stones, position of the stone in the kidney, kind of ureteroscope used, operative time measured from the beginning of the cystoscopy to withdrawal of all endoscopic equipments and from start to finish the insertion of the flexible ureteroscope into the kidney, lithotripsy technique (basketing without fragmentation, dusting or combined technique), endoscopic inspection at the end and presence of residual fragments > 2 mm in postoperative CT, composition of urinary calculi, 2 blood and urinary metabolic evaluations of each patient to be made between 45 and 90 days of the procedure, including: total calcium, parathyroid hormone (PTH), uric acid, urea, creatinine, venous blood gas, urine pH, urine culture, 24 hours urine dosage of calcium, sodium, citrate, oxalate, cystine, creatinine, urea, uric acid and phosphate. Other authors (8) demonstrated in a retrospective study that the size of the stone (p < 0.001), location (p< 0.001), multiplicity (p = 0.003), surgical time (p = 0.008) and exclusive use of flexible ureteroscope (p = 0.029) are associated with the presence of residual fragments.

Sensitivity and specificity of the combination US + Rx for identification of residual fragments on postoperative CT, predictive parameters for the best accuracy of the combination US + Rx and endoscopic end inspection and the occurence of complications such as ureteral lesion, renal dilatation, visits to the emergency room for pain control, need for additional procedures are going to be determined.

Statistics

The comparison between the methods of assessment of residual fragments will be done with Cochran test and prediction of parameters to avoid CT will be made with multiple logistic regression, using the IPSS 16.0 program, with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Kidney calculi > 5 mm and < 20 mm or < 15 mm in lower kidney calyx

Exclusion Criteria:

* Patients with kidney malformations, ureteral stenosis, previous ipsilateral kidney surgery, hydronephrosis, indwelling double J stent and contraindications for URF are going to be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic renal calculi
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
residual calculi > 2mm by CT | 90 days

SECONDARY OUTCOMES:
complications by CT | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Danilovic, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided